CLINICAL TRIAL: NCT05636046
Title: Transseptal Catheterization Registry. An Italian Overview
Brief Title: Transseptal Italian Registry (TITLE)
Acronym: TITLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Luigi Sacco University Hospital (Other)
Responsible Party: Principal Investigator, Gianfranco Mitacchione, Principal Investigator - Cardiac Electrophysiologist, Luigi Sacco University Hospital
Other Study IDs: TITLE-registry
Record Dates: First submitted 2022-11-20; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Arrhythmia; Cardiac Disease
Keywords: Catheter ablation; Transseptal catheterization
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- transseptal catheterization performed without auxiliary tools: patients in whom transseptal catheterization have been performed without auxiliary tools
  Interventions: Procedure: transseptal catheterization
- transseptal catheterization performed with auxiliary tools: patients in who transseptal catheterization have been performed with the use of auxiliary tools
  Interventions: Procedure: transseptal catheterization

INTERVENTIONS:
Procedure: transseptal catheterization — puncture of interatrial septum at the level of fossa ovalis, using transseptal needle.
  Other Names: transseptal puncture

SUMMARY:
The goal of this observational study is to learn about the changing over the time of transseptal (TSP) catheterization for catheter ablation of arrhythmias in the left heart. This study aims to investigate if auxiliary tools for TSP catheterization improved the safety and efficacy.

DETAILED DESCRIPTION:
Data regarding transseptal catheterization in the Centers involved will be retrospectively collected over the past 10 years.

Will be collected:

1) patients characteristics

1. type of procedure requiring transseptal catheterization
2. success rate
3. adverse events
4. use of tools for transseptal catheterization:

   * intracardiac echocardiography (ICE) guidance
   * simplified transseptal puncture
   * "pig tail" catheter
   * "safe sept" guidewire
   * powered radiofrequency transseptal needle

ELIGIBILITY:
Inclusion Criteria:

* patients underwent transseptal catheterization of left side heart interventional procedures (catheter ablation)

Exclusion Criteria:

* patients with learning disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients underwent trasseptal catheterization for catheter ablation of arrhythmias in the left heart
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-11-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Adverse events related to inadvertent puncture cardiac structures other than atrial septum | Procedure time
  absence of adverse events related to transseptal catheterization
Accomplishment of transseptal catheterization and electrophysiology procedure requiring transseptal catheterization | Procedure time
  accomplishment fo transseptal catheterization

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Presidio Ospedaliero G. Salesi, Ancona
  - Ospedale Policlinico Sant'Orsola-Malpighi, Bologna
  - Spedali Civili di Brescia, Brescia
  - Ospedale Desenzano del Garda, Desenzano del Garda
  - Centro Cardiologico Monzino, Milan
  - Luigi Sacco University Hospital, Milan
  - Ospedale San Raffaele, Milan
  - Ospedale San Gerardo, Monza
  - Ospedale Policlinico Universitario Agostino Gemelli, Roma
  - Ospedale Di Circolo e Fondazione Macchi, Varese

IPD SHARING:
Plan to Share IPD: No